CLINICAL TRIAL: NCT06060782
Title: Clinical Study on the Efficacy and Safety of Auto-HSCT in Adult Patients with Burkitt Lymphoma, Lymphoblastic Lymphoma, and Acute Lymphoblastic Leukemia Who Received TCCA Conditioning Regimen
Brief Title: Thiotepa, Cyclophosphamide, Clarithromycin and Cytarabine
Acronym: TCCA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZDWY.XYZLK.002
Record Dates: First submitted 2023-09-25; First posted 2023-09-29 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Burkitt Lymphoma; Lymphoblastic Lymphoma, Adult; Acute Lymphoblastic Leukemia, Adult
Keywords: Thiotepa; Cyclophosphamide; Cladribine; Cytarabine; conditioning regimen
MeSH Terms: conditions — Burkitt Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Thiotepa; Cyclophosphamide; Cladribine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- subject group (Experimental)
  Interventions: Drug: Thiotepa, cyclophosphamide, cladribine, and cytarabine conditioning regimen

INTERVENTIONS:
Drug: Thiotepa, cyclophosphamide, cladribine, and cytarabine conditioning regimen — All enrolled patients received TCCA conditioning regimen（） before auto-HSCT:
  Thiotepa 5mg/kg, -8, -7 days Cyclophosphamide 40mg/kg, -6, -5 days Cladribine 5mg/m2, -4, -3, -2 days Cytarabine 2g/m2, -4, -3, -2 days
  Other Names: TCCA conditioning regimen group

SUMMARY:
This study is an observational study on the efficacy and safety of auto-HSCT in adult patients with Burkitt lymphoma, lymphoblastic lymphoma, and acute lymphoblastic leukemia who received TCCA conditioning regimen. The study plans to include 28 patients who received the TCCA regimen for pre-transplantation pretreatment before auto-HSCT. Maintenance treatment will be carried out after transplantation for 1 year to observe the efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily sign the informed consent form, which must be signed by the patient himself.

  2. ALL patients confirmed by bone marrow cell morphology, immunology, and genetics; 3. PH+ALL patients who achieve s3CMR (definition: achieve molecular biological remission in the early stage of initial treatment (within 3 months) and maintain remission); 4. Ph-B-ALL patients who have reached MRD- after 3 courses of chemotherapy and continue to be MRD-; adult patients with Burkitt lymphoma and lymphoblastic lymphoma confirmed by histopathology and molecular genetics; 5. Adult patients with Burkitt lymphoma and lymphoblastoma, if the bone marrow is not involved, can achieve PR or above after induction; if the bone marrow is involved at the time of initial diagnosis, 3 courses of chemotherapy are required to reach MRD- and continue to be MRD-.

  6. Patients receiving autologous hematopoietic stem cell transplantation (auto-HSCT); 7. Age ≥18 years and ≤65 years old, male or female; 8. Eastern Cooperative Oncology Group Performance Status (ECOG-PS) score of 0-2;

Exclusion Criteria:

* 1. Have a history of cancer and have received any treatment for this tumor in the past 3 years, except for superficial bladder cancer, basal cell or squamous cell carcinoma of the skin, cervical intraepithelial carcinoma (CIN), or prostate epithelium Internal carcinogenesis (PIN); 2. Known to be serologically positive for HIV, active hepatitis B, active hepatitis C virus or syphilis; 3. Suffering from mental illness or other conditions and unable to cooperate with the requirements of research treatment and monitoring; 4. Pregnant patients or patients who cannot take appropriate contraceptive measures during treatment; 5. Received hematopoietic stem cell transplantation within the past 1 year; 6. Active heart disease, defined as one or more of the following:

  1. Have a history of uncontrolled or symptomatic angina;
  2. Myocardial infarction less than 6 months from study enrollment;
  3. Have a history of arrhythmia that requires drug treatment or has severe clinical symptoms;
  4. Uncontrolled or symptomatic congestive heart failure (>NYHA class 2);
  5. The ejection fraction is lower than the lower limit of the normal range. 7. Patients who meet the following criteria:

  <!-- -->

  1. Major surgery (except diagnostic surgery) is planned within 4 weeks before enrollment or during the study period, or the surgical wound has not fully healed before enrollment;
  2. Those who have received (attenuated) live vaccines within 4 weeks before enrollment;
  3. Patients with suspected active or latent tuberculosis;
  4. Participate in other clinical trials one month before enrollment 8. Those who the researcher believes are not suitable for enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
3-year recurrence-free survival rate | 3 years after transplantation

SECONDARY OUTCOMES:
3-year overall survival rate | 3 years after transplantation
3-year recurrence rate | 3 years after transplantation
Transplant-related mortality | From the beginning of conditioning to 3 years after transplantation
The patient's tolerance and mucositis grade | From the beginning of conditioning chemotherapy to hematopoietic reconstitution
The incidence of cataracts and second tumors | From the beginning of conditioning to 3 years after transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided